CLINICAL TRIAL: NCT00551044
Title: Bicalutamide Monotherapy Preserves Bone Mineral Density, Muscle Strength and Has Significant Quality of Life Benefits for Men With Advanced Prostate Cancer
Brief Title: Bicalutamide Monotherapy Has Significant Quality of Life Benefits for Men With Advanced Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wirral University Teaching Hospital NHS Trust (Other)
Collaborators: AstraZeneca (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 96/02
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Last update posted 2007-10-30 (Estimated); Status verified 2007-08

CONDITIONS: Prostatic Neoplasms
Keywords: prostatic neoplasms; bicalutamide; quality of life; osteoporosis
MeSH Terms: conditions — Prostatic Neoplasms; Osteoporosis | interventions — bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bicalutamide (Active Comparator): Osteoporotic patients (T score ≤ -2.5) on bicalutamide
  Interventions: Drug: Bicalutamide

INTERVENTIONS:
Drug: Bicalutamide — Bicalutamide 150mg once daily, oral administration, for 12 months

SUMMARY:
The aim of this study is to comprehensively monitor the effects of a nonsteroidal antiandrogen in patients requiring hormone manipulation for prostate cancer

DETAILED DESCRIPTION:
Androgen deprivation therapy is the mainstay of treatment for advanced prostate cancer. There is an increasing tendency towards earlier treatment with hormone manipulation. However, luteinizing hormone-releasing agonists decrease serum testosterone to castrate levels within two weeks of commencement.They are associated with loss of libido, loss of muscle bulk and accelerated bone loss. Osteoporotic patients are at high risk of fragility fractures. An alternative is the nonsteroidal antiandrogen bicalutamide which blocks testosterone at the receptor level, allowing androgen deprivation in the prostate without reducing circulating levels of testosterone. This should preserve the desired effects on other androgen-sensitive tissue, resulting in an advantageous side effect profile. The aim of our study is to closely monitor osteoporotic patients commencing bicalutamide for a period of 12 months. Patients will be reviewed in a dedicated prostate cancer clinic every 3 months. Patients will be questioned regarding adverse events. Renal and liver function tests, prostate specific antigen, testosterone, estradiol and bone turnover markers will be measured 3 monthly. Measurement of height , weight, body mass index, quadriceps strength using dynamometry, and skeletal mass using arm anthropometry (mid-arm circumference and triceps skinfold thickness), will be carried out 3 monthly. Quality of life issues will be assessed 3 monthly using the Rand 36-Item Health Survey (SF36) and University of California-Los Angeles Prostate Cancer Index (UCLAPCI). Patients will undergo bone densitometry of the forearm at baseline and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Osteoporotic patients (T score ≤ -2.5) with advanced prostate cancer requiring hormone manipulation, due to biochemical relapse following either radical prostatectomy, radiotherapy, brachytherapy, or biochemical progression after initially being observed with prostate cancer.

Exclusion Criteria:

* Severe hepatic insufficiency, with bilirubin above reference range
* Previous systemic therapy for prostate cancer
* Radiotherapy within 6 months
* Previous other invasive malignancies
* Any severe concomitant disease.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2003-08; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Quality of life (using Rand 36-Item Health Survey SF-36) | 3 monthly for 1 year

SECONDARY OUTCOMES:
Renal & liver function tests, PSA, testosterone, estradiol | 3 monthly for 1 year
Body Mass Index, arm anthropometry (mid-upper arm circumference and triceps skin fold thickness), dynamometry (quadriceps muscle strength) | 3 monthly for 1 year
Bone turnover markers (bone-specific alkaline phosphatase, N-terminal propeptide of type I collagen, C-telopeptide crosslinks of type I collagen, urine N-telopeptide of tyoe I collagen corrected for creatinine | 3 monthly for 12 months
Peripheral bone densitometry of non-dominant forearm | At baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nigel J Parr, MBBS, FRCS(Urol), MD, Principal Investigator — Wirral University Teaching Hospital NHS Trust
Locations (1):
- Wirral University Teaching Hospitals NHS Trust, Upton, Wirral, Merseyside, United Kingdom

REFERENCES:
- [Derived] Wadhwa VK, Weston R, Parr NJ. Bicalutamide monotherapy preserves bone mineral density, muscle strength and has significant health-related quality of life benefits for osteoporotic men with prostate cancer. BJU Int. 2011 Jun;107(12):1923-9. doi: 10.1111/j.1464-410X.2010.09726.x. Epub 2010 Oct 15. PMID 20950306